CLINICAL TRIAL: NCT02430987
Title: Prevalence of Hypoactive Sexual Desire Disorder in Sexually Active Postmenopausal Women With Metabolic Syndrome Women Attending in a Public Hospital Clinic in Brazil: a Cross-sectional Study
Brief Title: Low Sexual Desire and Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 40594814.4.0000.5479
Record Dates: First submitted 2015-04-27; First posted 2015-04-30 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Menopause; Metabolic Syndrome; Hypoactive Sexual Desire Disorder; Obesity; Sexual Dysfunction
Keywords: menopause; hypoative sexual desire disorder; metabolic syndrome; obesity
MeSH Terms: conditions — Metabolic Syndrome; Sexual Dysfunctions, Psychological; Obesity; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metabolic syndrome (Active Comparator): The MetS diagnosis was determined by following the guidelines defined by the Adult Treatment Panel (ATP III) (8): (1) Abdominal circumference (AC) ?88cm; (2) HDL-cholesterol < 50mg/dL; (3) triglycerides > 150mg/dL; (4) arterial blood pressure (SAH) > 130/85mmHg; and (5) fasting glucose > 110mg/dL. The women considered as carrying MetS were those with at least three of the components described.
  Sexual function was assessed by completion of the Female Sexual Function Index (FSFI), a questionnaire validated for Brazilian Portuguese
  Interventions: Diagnostic Test: Female sexual function index questionnaire; Diagnostic Test: Evaluation of presence of metabolic syndrome
- Obesity (Placebo Comparator): women were stratified into 3 groups by body mass index (BMI): Group 1: BMI of 18.5 to 24.9kg/m2 (Normal BMI Group), Group 2: BMI of 25 to 29.9kg/m2 (Overweight Group); Group 3: BMI of 30kg/m2 to 34.5kg/m2 or higher) (Obese Group Sexual function was assessed by completion of the Female Sexual Function Index (FSFI), a questionnaire validated for Brazilian Portuguese
  Interventions: Diagnostic Test: Female sexual function index questionnaire; Diagnostic Test: Evaluation of presence of metabolic syndrome; Diagnostic Test: Evaluation of the body mass index

INTERVENTIONS:
Diagnostic Test: Female sexual function index questionnaire — Sexual function was assessed by completion of the Female Sexual Function Index (FSFI), a questionnaire validated for Brazilian Portuguese with 19 items measuring female sexual function. Cut-off points of >23 and > 26.5 were adopted to define a diagnosis of Female Sexual Function based on the Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM -IV- TR) by the American Psychiatric Association, duration criteria > 24 weeks.
  A score of 5 or less on the combination of items comprising the desire domain of the FSFI questionnaire was used to define the diagnosis of Hypoactive Sexual Desire Disorder (HSDD) in postmenopausal women We consider that a score of 6 or more the woman does not present with HSDD.
  Other Names: diagnostic of sexual dysfunction; diagnostic of hypoactive sexual desire disorder
Diagnostic Test: Evaluation of presence of metabolic syndrome — The MetS diagnosis was determined by following the guidelines defined by the Adult Treatment Panel (ATP III) (8): (1) Abdominal circumference (AC) ?88cm; (2) HDL-cholesterol < 50mg/dL; (3) triglycerides > 150mg/dL; (4) arterial blood pressure (SAH) > 130/85mmHg; and (5) fasting glucose > 110mg/dL. The women considered as carrying MetS were those with at least three of the components described.
Diagnostic Test: Evaluation of the body mass index — women were stratified into 3 groups by body mass index (BMI): Group 1: BMI of 18.5 to 24.9kg/m2 (Normal BMI Group), Group 2: BMI of 25 to 29.9kg/m2 (Overweight Group); Group 3: BMI of 30kg/m2 to 34.5kg/m2 or higher) (Obese Group
  Other Names: Diagnosis of obesity
  Arms: Obesity

SUMMARY:
Objective: To evaluate the prevalence of hypoactive sexual desire disorder (HSDD) in postmenopausal women diagnosed with metabolic syndrome (MS) and to compare it to that of a control group without MS.

Design: Cross-sectional study. Setting: Two public tertiary hospitals in the state of São Paulo, Brazil. Population: Two-hundred ninety-one postmenopausal women between 40 and 65 years of age.

Methods: Sexual function was evaluated using the Female Sexual Function Index (FSFI) questionnaire and DSM-IV-TR diagnostic criteria and was related to the diagnosis of MS, which was determined according to the guidelines defined by the Adult Treatment Panel (ATP III).

Main outcome measures: Analysis of sexual function with emphasis on sexual desire (HSDD), the presence of MS and its components.

DETAILED DESCRIPTION:
Study location Menopause Outpatient Clinic of the School of Medical Sciences of Santa Casa de São Paulo (FCMSCSP) and the 'Leonor Mendes de Barros' Maternity Hospital (HMLMB).

Population From 2015 to 2018, we were invited 1,200 postmenopausal women who regularly visit these institutions to undergo routine climacteric screening. After applying the inclusion and exclusion criteria, 291 sexually actives women were selected and invited to participate in the study. All participants signed an informed consent form.

Design A cross-sectional study was conducted. After the women agreed to participate in the study, they were stratified into 2 groups: group 1 - patients with MS and group 2 - control (without MS); the women in each group had diagnoses of HSDD and FSD. The results for women in group 1 were compared with those for women without MS in group 2.

Main outcome measures

Sexual function was assessed using the Female Sexual Function Index (FSFI) questionnaire,8 validated for the Portuguese language9 with 19 items that measure female sexual function. Cut-off points of > 2310 and > 26.58 were adopted to define the presence of FSD. A score of 5 or less for the sum of items that compose the desire domain of the FSFI questionnaire was used to define the presence of HSDD in postmenopausal women.11 The questions are as follows:

How often do you feel sexual desire or interest? 5 = Almost always or always 4 = Most times (more than half the time) 3 = Sometimes (about half the time) 2 = A few times (less than half the time) 1 = Almost never or never How would you rate your level of sexual desire or interest? 5 = Very high 4 = High 3 = Moderate 2 = Low

1 = Very low or none at all We considered that a woman with a score of 6 or higher did not have HSDD. The diagnosis of FSD was based on the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) by the American Psychiatric Association.

The diagnosis of sexual dysfunction was established by an experienced sexologist (GMDS) trained in the diagnosis of FSD using the FSFI. The women provided their responses in a private room. The Beck Inventory12 was used to rule out depression in patients with a history of the disease/distress (score >14).

The diagnosis of MS was determined following the guidelines defined by the Adult Treatment Panel: waist circumference (WC) > 88 cm; high-density lipoprotein (HDL)-cholesterol ≤ 50 mg/dL; triglycerides ≥ 150 mg/dL; blood pressure (BP) ≥ 130/85 mmHg; and fasting glucose level ≥ 110 mg/dL. The use of medication and/or a previous diagnosis of the condition did not exclude the use of a component for the diagnosis of MS.

A semi-structured questionnaire was applied to each participant to collect demographic, socioeconomic, and clinical information. BP, WC and body mass index (BMI) were measured. Next, a gynaecological exam was performed, and a cytology sample was collected for a Pap smear.

Laboratory tests were conducted (total cholesterol and fractions, triglycerides and fasting glucose), along with bilateral mammography and transvaginal ultrasound exams, according to the routine procedures of the department.

The study was conducted in accordance with the protocol and the principles established in the Declaration of Helsinki (1996), the International Conference on Harmonization Harmonized Tripartite Guideline: Good Clinical Practice Guidelines, and regulatory requirements. The protocol was approved by the Human Research Ethics Committee of the School of Medical Sciences of the Santa Casa de São Paulo Hospital and the 'Leonor Mendes de Barros' Maternity Hospital (CAAE number 40594814.4.0000.5479) and registered as a clinical trials under ID NCT02430987.

The inclusion criteria were as follows:

* 40-65 years of age;
* One year of amenorrhea and FSH > 30 mIU/mL14;
* Sexually active - women with regular sexual activity and to have penetrative sex with a partner without a history of sexual dysfunction in the last 4 weeks; and
* Use of oestrogen and progesterone oral or parenteral for over 6 months. This item is to prevent hot flashes and vaginal dryness interference in sexual function.

The exclusion criteria were as follows:

* Women in the menopause transition period and/or with FSH <30 mIU/mL;
* Sexually inactive;
* Partner with history of sexual dysfunction, such as erectile dysfunction and/or premature ejaculation;
* Any other form of sexual dysfunction or any other psychiatric disorder that may affect sexual function;
* Diagnosis of depression, with a score of > 14 on Beck's Depression Inventory;
* Use of oestrogen and progesterone oral or parenteral prescribed less than 6 months ago or prescribed for low sexual desire (tibolone);
* Use of drugs that, according to the examiner's evaluation, may affect sexual function;
* History of bilateral oophorectomy; and
* Diagnosed with cancer (breast, cervix, endometrium, ovary, intestines, among others);

Data analysis To analyse the sample, the characteristics of the women participating in the study were described using absolute and relative frequencies for qualitative measures and summary measures (mean, standard deviation, median, minimum and maximum) for quantitative measurements.

With the objective of analysing the relationships between the population characteristics and the FSFI questionnaire domains, generalized linear models with a gamma distribution and identity link function were created to compare the scores according to the categories of interest adjusted for age, education level, race/colour, marital status and religion.

The FSFI questionnaire scores were described based on the presence or absence of MS and compared using the Mann-Whitney test. The analyses were performed using IBM-SPSS software for Windows version 20.0 (IBM, IL, Chicago, USA). Microsoft Excel 2003 software was used to store the data and results, and the statistical package StatistiXL (Statistical Power for MS Excel version 1.8, 2007) was used for the statistical analyses. The tests were performed with a significance level of 5%.

The sample size calculation was based on a confidence level (1-alpha) = 95, a power (% of probability of detection) = 80, a ratio of controls to cases = 1, a hypothetical proportion of controls with exposure = 40, a hypothetical proportion of cases with exposure = 57.14, and a least extreme odds ratio to be detected = 2.00, resulting in a sample size totalling 288 patients (144 cases and 144 controls).

ELIGIBILITY:
The inclusion criteria were as follows:

* 40-65 years of age;
* One year of amenorrhea and FSH > 30 mIU/mL14;
* Sexually active - women with regular sexual activity and to have penetrative sex with a partner without a history of sexual dysfunction in the last 4 weeks; and
* Use of oestrogen and progesterone oral or parenteral for over 6 months. This item is to prevent hot flashes and vaginal dryness interference in sexual function.

The exclusion criteria were as follows:

* Women in the menopause transition period and/or with FSH <30 mIU/mL;
* Sexually inactive;
* Partner with history of sexual dysfunction, such as erectile dysfunction and/or premature ejaculation;
* Any other form of sexual dysfunction or any other psychiatric disorder that may affect sexual function;
* Diagnosis of depression, with a score of > 14 on Beck's Depression Inventory;
* Use of oestrogen and progesterone oral or parenteral prescribed less than 6 months ago or prescribed for low sexual desire (tibolone);
* Use of drugs that, according to the examiner's evaluation, may affect sexual function;
* History of bilateral oophorectomy; and
* Diagnosed with cancer (breast, cervix, endometrium, ovary, intestines, among others);

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 291 (Actual)
Dates: Start 2014-09; Primary Completion 2018-04 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
application of questionnaire | 1 year
  application of questionnaire about sexuality and sexual function

SECONDARY OUTCOMES:
Body mass index | 2 years
  Evaluated the body mass index of all participants
Metabolic syndrome | 3 years
  Evaluated the diagnosis of metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Maximiliano Dutra da Silva, PhD, Principal Investigator — Faculdade de Ciências Médicas da Santa Casa de São Paulo
Locations (1):
- Rua Maria José Pomar, 322 Apartamento 172 C, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Silva GM, Lima SM, Moraes JC. [Evaluation of sexual function in postmenopause women with metabolic syndrome]. Rev Bras Ginecol Obstet. 2013 Jul;35(7):301-8. doi: 10.1590/s0100-72032013000700004. Portuguese. PMID 24080842
- [Result] Silva GMDD, Lima SMRR, Reis BFD, Macruz CF, Postigo S. Evaluation of Obesity Influence in the Sexual Function of Postmenopausal Women: A Cross-Sectional Study. Rev Bras Ginecol Obstet. 2019 Nov;41(11):660-667. doi: 10.1055/s-0039-1700795. Epub 2019 Nov 19. PMID 31745959
- [Derived] Dutra da Silva GM, Rolim Rosa Lima SM, Reis BF, Macruz CF, Postigo S. Prevalence of Hypoactive Sexual Desire Disorder Among Sexually Active Postmenopausal Women With Metabolic Syndrome at a Public Hospital Clinic in Brazil: A Cross-sectional Study. Sex Med. 2020 Sep;8(3):545-553. doi: 10.1016/j.esxm.2020.05.008. Epub 2020 Jun 24. PMID 32593675